CLINICAL TRIAL: NCT06779474
Title: Laparoscopic Associating Liver Partition With Portal Vein Ligation for Staged Hepatectomy (ALPPS) for Colorectal Liver Metastases (CRLM)
Status: Not yet recruiting | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Director, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2022ZSLYEC-130
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Liver Metastases
Keywords: Colorectal liver metastases; Associating liver partition and portal vein ligation for staged hepatectomy; Laparoscopic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Laparoscopic ALPPS group: CRLM patients with insufficient future liver remnant who are performed laparoscopic associating liver partition with portal vein ligation for staged hepatectomy
  Interventions: Procedure: Laparoscopic ALPPS

INTERVENTIONS:
Procedure: Laparoscopic ALPPS — Laparoscopic Associating Liver Partition With Portal Vein Ligation for Staged Hepatectomy

SUMMARY:
Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) is a procedure used for patients with initially unresectable colorectal liver metastases (CRLM). However, the procedure has been reported to be associated with high morbidity and mortality. Laparoscopic ALPPS has recently been reported as a minimally invasive technique that reduces perioperative risks. This study aimed to assess the safety and feasibility of full laparoscopic ALPPS in patients with CRLM.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years < 75 of age.
2. ECOG performance status 0-1.
3. Histologically confirmed colorectal adenocarcinoma.
4. Imaging (CT or MRI) or pathological confirmation of liver metastasis.
5. Child-Pugh grade A liver function.
6. FLR/sTLV (standardized total liver volume) < 30% (patients without underlying liver diseases)or < 40% (patients with liver diseases, such as hepatic steatosis, cirrhosis, or liver damage after chemotherapy).
7. The indication of surgery is evaluated by a multidisciplinary team attended by hepatobiliary surgeons, oncologists, hepatologists and radiologists.

Exclusion Criteria:

1. Patients with unresectable extrahepatic metastatic disease (except potentially resectable lung metastases) or primary tumor.
2. Patients with severe concomitant diseases who are intolerance of major liver surgery by the judgment of the surgeon.
3. Diagnosis of other malignant tumors within the past 5 years.
4. Intention to become pregnant during the course of the study.
5. Inability to comply with the study protocol.
6. Previous enrollment in the current study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are hospitalized at the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | within the first 90 days after the first stage of ALPPS
  Morbidity and mortality of laparoscopic ALPPS

SECONDARY OUTCOMES:
Resection rate | within the first 14 days after the second stage of ALPPS
  R0 resection rate of laparoscopic ALPPS
Survival | 3 years
  follow-up after the surgery every 3 months, to evaluate recurrence, death, analysis 1-year, 3-year overall survival rates，disease-free survival rates and recurrence rate.
Future liver remnant after surgery | 3 months
  Future liver remnant volume calculated 3 months after the stage 2 surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol